Novel Use of Cyclosporine Ophthalmic Emulsion 0.05% in a PROSE Device

NCT#: NCT04918823

Version: 8/27/2024

| v |
|---|

## Statistical Analysis

Statistical analysis was performed using Visual Studio Code (Microsoft Corp., Redmond WA) with python version 3.9.12. Subject data post-treatment was compared to their baseline data, collected prior to initiating use of the study drug. For Group A, the data collected at Visit 1A was considered to be their baseline data pre-intervention. For Group B, the data collected at Visit 1B was considered to be their baseline data (post-initiation of Purilens and pre-initiation of cyclosporine). The core algorithm used was based on statistical functions module scipy.stats. For univariate data analysis (before/after visits), paired t-test was performed since every patient received treatment. Paired t-test was conducted by scipy.stats. t test\_rel and <a href="https://www.statskingdom.com/paired-t-test-calculator.html">https://www.statskingdom.com/paired-t-test-calculator.html</a>. For bi-variate data, two-way ANOVA (Analysis of variance) was performed. Two-way ANOVA was conducted by sm. stats. anova\_lm(model) function. The significance level was set to a P-value of <0.05 in all instances of analysis.

